CLINICAL TRIAL: NCT04821713
Title: ENerGetics in Old AGE (ENGAGE Study) - Validation of Multiple Accelerometers and Physical Activity Questionnaires Against Indirect Calorimetry Under Laboratory and Free-living Conditions in Very Old Adults
Brief Title: Validation of Objectively and Subjectively Measured Physical Activity Against Energy Expenditure in Older Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); National Institutes of Health (NIH) (NIH); Maastricht University (Other); University of Wisconsin, Madison (Other); University of California, Berkeley (Other); University of Ulster (Other); University Ramon Llull (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paolo Caserotti, Professor, University of Southern Denmark
Other Study IDs: 65838; 5R01CA183570-05 (NIH)
Record Dates: First submitted 2021-03-01; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: no Condition, Community-dwelling 80+ Older Adults
Keywords: Accelerometer; Physical Activity; Sedentary behavior; Energy Expenditure; Older Adults
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine, saliva, plasms, serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Physical inactivity is identified as one of the most important modifiable risk factors for chronic diseases, functional loss and disability and reliable assessment tools of physical activity are crucial in both research and clinical settings.

Traditionally, physical activity and sedentary behavior have been primarily assessed with questionnaires. Recently, accelerometers have been widely used to measure physical activity, sedentary behavior and sleep patterns in ageing. Still, the diversity of brands and models, various assessment protocols (e.g. anatomic locations, sampling frequency), data processing and outcome measures have posed challenges to the interpretation and comparability of results across studies. Therefore, despite some limitations, questionnaires are still considered an important assessment method, especially in large-scale studies. In order to bridge the differences in the interpretation of data from questionnaires to accelerometers among older adults, there is a need to validate existing physical activity and sedentary behavior questionnaires with energy expenditure in this population.

Energy expenditure has been used to "translate" accelerometer output into physiological outcomes. Nevertheless, several issues remain unresolved, including (1) limited calibration studies focusing on older adults; (2) resting metabolic rate and maximum physiological capacity typically decrease with aging, which makes daily activities "more intense" for an older person compared to a younger person; and (3) the same accelerometer metric measured at different body positions may be linked to completely different physiological outcomes.

Such diverse physiological impact according to the anatomical placement of accelerometers requires a rigorous harmonization of metrics from the accelerometers with energy expenditure during representative activities at different intensities.

The aims of this methodological study focusing on 80+ year-olds are to:

1. develop cut-points from accelerometers at different anatomical positions for different intensities of physical activity based on energy expenditure during semi-standardized daily tasks in the lab.
2. validate accelerometer at different anatomical positions against energy expenditure measured by double-labelled water (DLW) in free-living conditions.
3. validate existing physical activity and sedentary behavior questionnaires against DLW in free-living conditions.

DETAILED DESCRIPTION:
Background

Physical inactivity has been estimated to cause 5.3 million deaths per year globally and is identified as one of the most important modifiable risk factors for chronic diseases, functional loss and disability. To correctly identify and study physical inactivity in old age, reliable assessment tools are crucial in both research and clinical settings.

Recent technological advancements in wearable activity monitors have led to a growing number of large, population-based studies using accelerometers to measure physical activity, sedentary behavior (in terms of overall volume, intensity and pattern), and sleep among older adults. However, the wide use of accelerometers also brings challenges when comparing the results across different studies that use different brands and models, various assessment protocols (e.g. anatomic locations, sampling frequency), data processing procedures and report different outcomes. Different accelerometer set-ups (i.e. brand, model, body position, initialization protocol, etc.) may challenge the interpretation of health-enhancing effect of physical activity and detrimental effect of sedentary behavior simply because of methodological issues.

Accelerometers measure acceleration, defined as the change in velocity over time (Δv/t), which quantifies the volume and intensity of movement. In addition, acceleration is a vector quantity with components of magnitude and direction, which can be used to identify the position of accelerometer in relation to gravity. Therefore, accelerometer could also be used to distinguish posture (e.g. sitting, standing, lying down) depending on the site of placement.

Since raw acceleration signals are difficult to interpret, they are typically "translated" by calibration studies to physiological outcomes (e.g. energy expenditure, oxygen consumption) or behavioral categories (e.g. sitting, walking, running). Through regression modelling, calibration studies often produce point estimates of energy expenditure from accelerometer counts or establish a range of accelerometer counts for different physical activity intensity levels. This range of accelerometer counts is referred to as "cut-points" for different intensities of physical activity.

Before the use of accelerometers, physical activity and sedentary behavior has been primarily assessed with questionnaires. Even as the scale of accelerometer studies are growing rapidly, questionnaires are still considered an important assessment method when assessing physical activity and sedentary behavior in large-scale studies. Some accelerometers and questionnaires have been validated by objectively measured energy expenditure. But for physical activity questionnaires, the validity against objective methods (e.g. accelerometry, heart rate monitor and double-labelled water) were found to be moderate at best and very few validation studies focused on older adults. In order to bridge and interpret data from questionnaires to accelerometers among older adults, there is a need to validate existing physical activity and sedentary behavior questionnaires with energy expenditure in this population.

Energy expenditure has earlier been used to validate accelerometers and physical activity questionnaires metrics. Nevertheless, several issues remain unsolved: (1) despite the correlation between these methods has been reported to be high in few studies, the agreement is generally low especially in populations with altered metabolic states such as obese and overweight individuals; (2) while the total volume of physical activity is a clear metric which is presumably positively correlated with total daily energy expenditure, intensity of physical activity in older adults may be affected by a number of physiological determinants such as cardiovascular and neuromuscular function, inflammation status and malnutrition. Resting metabolic rate (RMR) and maximum physiological capacity (e.g. maximum oxygen update (VO2 max) typically decrease with age, which may be particular important as the same daily activities would likely be "more intense" to an older person compared to a younger person; (3) despite that numerous activity monitors provide similar metrics (e.g. counts/minutes), the physiological implication can be highly different depending on what such metrics stand for. For example, despite the output from accelerometers placed on wrist and on the hip may be identical (counts/minutes), the different magnitude of acceleration may have a completely different physiological relationship when assessed by physiological metrics (e.g. energy, oxygen uptake). Such diverse physiological impact according to the anatomical placement of accelerometers requires a rigorous harmonization of metrics from the accelerometers coupled with energy expenditure in representative activities at different intensities.

To date, validation studies with accelerometers worn on multiple body positions are scarce and not all studies uses energy expenditure as the reference. One way to disentangle the physiological meaning of physical activity and sedentary behavior is to anchor accelerometer output to objective measurements of physiological capacity such as VO2 max, oxygen uptake during semi-standardized activities performed at self-selected pace and overall energy expenditure during free-living conditions collected over a representative period of time. This will contribute to a deeper understanding and accurate interpretation of the accelerometer data among community-dwelling older adults and to provide more specific accelerometry-based recommendations for physical activity, especially for the oldest population.

Objectives

The aims of this methodological study are to:

1. develop hip-, wrist-, thigh-, and low back- worn accelerometer cut-points for different intensities of physical activity based on energy expenditure during semi-standardized daily tasks for the 80+ year-olds.
2. validate accelerometry at the wrist, hip, thigh, and low back for estimating energy expenditure in free-living conditions, measured by the gold standard of energy expenditure, double-labelled water (DLW).
3. validate existing physical activity and sedentary behavior questionnaires against gold standard of energy expenditure (DLW) in free-living conditions in the 80+ year-olds.

Recruitment and data collection procedures

The investigators will conduct a cross-sectional study with two modes of data collection: 1) in the laboratory; and 2) in the field. Participants will be recruited through two pathways: 1)(Pathway A) invited personally during the routine preventive home-visits performed by the Municipality of Odense ; (Pathway B)or 2) invited through a letter to community-dwelling older citizens who lives in the Municipality of Odense. Those who show interest to participate will then receive detailed written information about the project and will be invited to a medical screening after signing an informed consent. The entire testing procedure will span across 14 days as urine samples for DLW method is needed on Day 1 and Day 14. In between, participants will be invited to attend one for lab test for measuring energy expenditure during semi-standardized functional tasks.

Statistical considerations and data management A detailed data management plan will be followed in the collection, entering, and analysis of data. In the laboratory examination day, all measurement devices will be synchronized before the measurement begins.

Sample size Assuming that different accelerometers can capture same physical activity behaviour, in a test for agreement between two raters using the Kappa statistic, a sample size of 95 subjects achieves 80% power to detect a true Kappa value of 0.70 when there are 3 categories with frequencies equal to 0.01, 0.20, and 0.79. (representing estimated percentage of time spent in moderate-to-vigorous activity, light activity, and sedentary behavior in this population). This power calculation is based on an alpha of 0.05.

Creation of a research biobank

A research biobank (blood, urine, and saliva samples) will be created for the described project. The blood samples will be destroyed no later than 5 years after the project is ending. Blood samples will be taking at the facilities of the University (SDU). An authorized nurse or biomedical laboratory scientist will be in charge of obtaining blood samples from the participants. The biobank will be stored at SDU. In total, 8 urine samples will be obtained from each participant during the entire project period. Urine samples will be frozen and sent to USA for analysis. The urine samples will be anonymized and stored in the research biobank until the end of the project, when the samples will be destroyed. A trained project personnel will be in charge of collecting urine samples from the subjects. In this protocol, University of Southern Denmark acts as the controller of the biological materials collected (urine samples). Data processing agreements will be made between SDU and the University of Wisconsin, USA; and between SDU and University of California, Berkeley. The US processor shall comply with Danish law governing protection of personal data.

Ethical considerations

The research activities of this study will be carried out in accordance with the Declaration of Helsinki. All subjects will receive the pamphlets from The National Committee on Health Research Ethics regarding personal rights when participating in a health research project and aspects to consider before deciding to participate. This study will involve older adults, who are considered vulnerable individuals. It is important to acknowledge and respect participants' autonomy, i.e., they have to be able to decide by themselves their participation in the study with the right to withdraw at any stage. Moreover, a communication strategy suitable for this population will be applied to prevent any risk of enhancing vulnerability and stigmatization of the older adults.

This project will generate valuable and novel knowledge about how do objectively measure physical activity measured by different accelerometers on the same individual correlate with energy expenditure among in +80-year-old community-dwelling citizens; and whether these patterns differ according to protein level. These knowledges that can be used to optimize and target the preventive and treatment strategies for malnourished older adults hence offer a benefit for the individual older adult and for the health care sector. Thus, the investigators believe that the benefits from the study is greater than the limited discomforts that may follow participation. Subjects are covered by the Danish Patient Insurance Association and can thus receive insurance of financial compensation in case any damage occurs while participating in the research project. This information will be given to participants both verbally and written (in the pamphlets from The National Committee on Health Research Ethics) during recruitment.

All personal data will become anonymized and handled with full confidentiality in compliance with the Personal Data Processing Act. The procedure of personal data processing will be reported to the Danish Data Protection Agency in University of Southern Denmark. In this study protocol, only the anonymized urine and saliva samples will be sent abroad for analysis (details described earlier) with no linkage to any other personal data (e.g. CPR number, address, telephone number etc..).

Participants will not receive any compensation for their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged 80+ years old.
* Have intact cognitive function, evaluated by a score ≥ 3 in the short form of the Mini- mental state evaluation (MMSE)14.
* Signed an informed letter of consent.

Exclusion Criteria:

* Have severe organic or mental disease as determined by history
* Have terminal cancer.
* Are on chemotherapy.
* Have a drug and/or alcohol abuse (>50 g alcohol a day).
* Have been prescribed new medication within 2 months with potential to alter metabolism.
* Are hospitalized or bed-ridden because they will not be able to perform any of the tasks in the laboratory and movement during the free-living activity would be limited.
* Those who need assistive devices (including wheelchair, cane, walkers etc..) for lab testing.
* Those who are unable to speak and read Danish because they will not be able to follow instructions in the laboratory and during the free-living conditions.

Min Age: 80 Years | Sex: All
Age Groups: Older Adult
Study Population: Community-dwelling men and women aged 80 and above.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Accelerometer-assessed physical activity in free-living condition | Through study completion, an average of 14 days
  Physical activity and sedentary behavior measured from accelerometers at multiple body locations in free-living condition. Raw accelerometer data will be processed in standard protocol and summarized in counts per minutes in vector magnitude.
Energy expenditure in free-living condition | Through study completion, an average of 14 days
  Oxygen uptake measured by doubly labelled water under free-living condition
Accelerometer-assessed physical activity in the lab | During lab measurement days up to 3 days
  Physical activity and sedentary behavior measured from accelerometers at multiple body locations in the lab. Raw accelerometer data will be processed in standard protocol and summarized in counts per minutes in vector magnitude.
Energy expenditure in the lab | During lab measurement days up to 3 days
  Oxygen uptake measured by indirect calorimetry in the lab

SECONDARY OUTCOMES:
Self-reported physical activity | During lab measurement days up to 1 day
  Measured by existing and ad hoc physical activity questionnaires: International Physical Activity Questionnaire--short form (IPAQ--short form), Physical Activity Scale for the Elderly (PASE).
  IPAQ-SF: IPAQ-SF is measuring PA across three domains: walking, moderate PA and vigorous PA. The total amount of PA is the sum of the three domains.
  * Minimum 0 MET-minutes/week
  * Maximum 19278 MET-minutes/week (truncated)
  PASE: The instrument is suitable for over 65 years old and comprised of self-reported occupational, household and leisure activities items over a one week period. PASE scores are calculated from weights and frequency values for each of 12 types of activity.
  * Minimum 0 PASE score
  * Maximum 400 (or more) PASE score
  Physical Activity Scale: The physical activity scale is a 24-hours measure and encompasses sleep, sedentary behavior, work, leisure time, and sports activity in one measure.
  * Minimum 25 MET-time/day
  * Maximum 150 MET-time/day
Self-reported sedentary behavior | During lab measurement days up to 1 day
  Measured by the Sedentary Behaviour Questionnaire (SBQ).
  SBQ: The SBQ measures time spent in sedentary behavior across different domains during weekdays and weekend days.
  * Minimum 0 hours
  * Maximum 24 hours
Protein level | Up to 4 days
  Measured by 4-day food diary, protein screener, biomarkers from blood
Muscle mass with DEXA scan | During lab measurement days up to 1 day
  Measured by DEXA scan
Muscle mass | Up to 4 days
  D3-creatine method
Handgrip Strength | During lab measurement days up to 1 day
  Handgrip strength measured by dynamometer in kg.
Lower extremity function | During lab measurement days up to 1 day
  Short Physical Performance Battery (SPPB), scores from 0 to 12, higher score indicating better function
Functional walking test | During lab measurement days up to 1 day
  Walking speed from 6-minutes walking test
Cardiovascular function | During lab measurement days up to 1 day
  VO2 max test

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Caserotti, PhD, Principal Investigator — Department of Sports and Clinical Biomechanics, University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
All personal data will become anonymized and handled with full confidentiality in compliance with the Personal Data Processing Act and GDPR. The procedure of personal data processing will be reported to the Danish Data Protection Agency (Datatilsynet) in University of Southern Denmark. In this study protocol, only the anonymized urine and saliva samples will be sent abroad for analysis (details described earlier) with no linkage to any other personal data (e.g. CPR number, address, telephone number etc..).

REFERENCES:
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Strath SJ, Kaminsky LA, Ainsworth BE, Ekelund U, Freedson PS, Gary RA, Richardson CR, Smith DT, Swartz AM; American Heart Association Physical Activity Committee of the Council on Lifestyle and Cardiometabolic Health and Cardiovascular, Exercise, Cardiac Rehabilitation and Prevention Committee of the Council on Clinical Cardiology, and Council. Guide to the assessment of physical activity: Clinical and research applications: a scientific statement from the American Heart Association. Circulation. 2013 Nov 12;128(20):2259-79. doi: 10.1161/01.cir.0000435708.67487.da. Epub 2013 Oct 14. PMID 24126387
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Worldwide trends in insufficient physical activity from 2001 to 2016: a pooled analysis of 358 population-based surveys with 1.9 million participants. Lancet Glob Health. 2018 Oct;6(10):e1077-e1086. doi: 10.1016/S2214-109X(18)30357-7. Epub 2018 Sep 4. PMID 30193830
- [Background] Freedson P, Pober D, Janz KF. Calibration of accelerometer output for children. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S523-30. doi: 10.1249/01.mss.0000185658.28284.ba. PMID 16294115
- [Background] Pisanu S, Deledda A, Loviselli A, Huybrechts I, Velluzzi F. Validity of Accelerometers for the Evaluation of Energy Expenditure in Obese and Overweight Individuals: A Systematic Review. J Nutr Metab. 2020 Aug 4;2020:2327017. doi: 10.1155/2020/2327017. eCollection 2020. PMID 32832147
- [Background] Doherty A, Jackson D, Hammerla N, Plotz T, Olivier P, Granat MH, White T, van Hees VT, Trenell MI, Owen CG, Preece SJ, Gillions R, Sheard S, Peakman T, Brage S, Wareham NJ. Large Scale Population Assessment of Physical Activity Using Wrist Worn Accelerometers: The UK Biobank Study. PLoS One. 2017 Feb 1;12(2):e0169649. doi: 10.1371/journal.pone.0169649. eCollection 2017. PMID 28146576
- [Background] Hoogendijk EO, Deeg DJ, Poppelaars J, van der Horst M, Broese van Groenou MI, Comijs HC, Pasman HR, van Schoor NM, Suanet B, Thomese F, van Tilburg TG, Visser M, Huisman M. The Longitudinal Aging Study Amsterdam: cohort update 2016 and major findings. Eur J Epidemiol. 2016 Sep;31(9):927-45. doi: 10.1007/s10654-016-0192-0. Epub 2016 Aug 20. PMID 27544533
- [Background] Arnardottir NY, Koster A, Van Domelen DR, Brychta RJ, Caserotti P, Eiriksdottir G, Sverrisdottir JE, Launer LJ, Gudnason V, Johannsson E, Harris TB, Chen KY, Sveinsson T. Objective measurements of daily physical activity patterns and sedentary behaviour in older adults: Age, Gene/Environment Susceptibility-Reykjavik Study. Age Ageing. 2013 Mar;42(2):222-9. doi: 10.1093/ageing/afs160. Epub 2012 Oct 31. PMID 23117467
- [Background] Crouter SE, Churilla JR, Bassett DR Jr. Estimating energy expenditure using accelerometers. Eur J Appl Physiol. 2006 Dec;98(6):601-12. doi: 10.1007/s00421-006-0307-5. Epub 2006 Oct 21. PMID 17058102
- [Background] Barnett A, van den Hoek D, Barnett D, Cerin E. Measuring moderate-intensity walking in older adults using the ActiGraph accelerometer. BMC Geriatr. 2016 Dec 8;16(1):211. doi: 10.1186/s12877-016-0380-5. PMID 27931188
- [Background] Matthew CE. Calibration of accelerometer output for adults. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S512-22. doi: 10.1249/01.mss.0000185659.11982.3d. PMID 16294114
- [Background] Koster A, Shiroma EJ, Caserotti P, Matthews CE, Chen KY, Glynn NW, Harris TB. Comparison of Sedentary Estimates between activPAL and Hip- and Wrist-Worn ActiGraph. Med Sci Sports Exerc. 2016 Aug;48(8):1514-1522. doi: 10.1249/MSS.0000000000000924. PMID 27031744
- [Background] Santos-Lozano A, Santin-Medeiros F, Cardon G, Torres-Luque G, Bailon R, Bergmeir C, Ruiz JR, Lucia A, Garatachea N. Actigraph GT3X: validation and determination of physical activity intensity cut points. Int J Sports Med. 2013 Nov;34(11):975-82. doi: 10.1055/s-0033-1337945. Epub 2013 May 22. PMID 23700330
- [Background] Sharifzadeh M, Bagheri M, Speakman JR, Djafarian K. Comparison of total and activity energy expenditure estimates from physical activity questionnaires and doubly labelled water: a systematic review and meta-analysis. Br J Nutr. 2021 May 14;125(9):983-997. doi: 10.1017/S0007114520003049. Epub 2020 Jul 28. PMID 32718378
- [Background] Helmerhorst HJ, Brage S, Warren J, Besson H, Ekelund U. A systematic review of reliability and objective criterion-related validity of physical activity questionnaires. Int J Behav Nutr Phys Act. 2012 Aug 31;9:103. doi: 10.1186/1479-5868-9-103. PMID 22938557
- [Background] Lewis LS, Hernon J, Clark A, Saxton JM. Validation of the IPAQ Against Different Accelerometer Cut-Points in Older Cancer Survivors and Adults at Risk of Cancer. J Aging Phys Act. 2018 Jan 1;26(1):34-40. doi: 10.1123/japa.2016-0207. Epub 2017 Dec 7. PMID 28422585
- [Background] Nishida Y, Tanaka S, Nakae S, Yamada Y, Morino K, Kondo K, Nishida K, Ohi A, Kurihara M, Sasaki M, Ugi S, Maegawa H, Ebine N, Sasaki S, Katsukawa F. Validity of the Use of a Triaxial Accelerometer and a Physical Activity Questionnaire for Estimating Total Energy Expenditure and Physical Activity Level among Elderly Patients with Type 2 Diabetes Mellitus: CLEVER-DM Study. Ann Nutr Metab. 2020;76(1):62-72. doi: 10.1159/000506223. Epub 2020 Mar 13. PMID 32172232
- [Derived] Skjodt M, Brond JC, Tully MA, Tsai LT, Koster A, Visser M, Caserotti P. Moderate and Vigorous Physical Activity Intensity Cut-Points for Hip-, Wrist-, Thigh-, and Lower Back Worn Accelerometer in Very Old Adults. Scand J Med Sci Sports. 2025 Jan;35(1):e70009. doi: 10.1111/sms.70009. PMID 39753998
- [Derived] Skjodt M, Tully MA, Tsai LT, Gejl KD, Ortenblad N, Jensen K, Koster A, Visser M, Andersen MS, Caserotti P. Need to Revise Classification of Physical Activity Intensity in Older Adults? The Use of Estimated METs, Measured METs, and V̇O2 Reserve. J Gerontol A Biol Sci Med Sci. 2024 Jul 1;79(7):glae120. doi: 10.1093/gerona/glae120. PMID 38703071